CLINICAL TRIAL: NCT01960777
Title: Chronic Pain After Inguinal Hernia Repair, ONSTEP vs. Laparoscopic Approach, A Randomised Observer Blinded Multicenter Study
Brief Title: Chronic Pain After Inguinal Hernia Repair, the ONSTEP Technique Versus the Laparoscopic Approach
Acronym: ONLAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jacob Rosenberg (Other)
Responsible Party: Sponsor-Investigator, Jacob Rosenberg, Professor, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ONLAP
Record Dates: First submitted 2013-10-09; First posted 2013-10-11 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Hernia, Inguinal; Chronic Pain
Keywords: Hernia, Inguinal; Laparoscopy; Onstep
MeSH Terms: conditions — Hernia, Inguinal; Chronic Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Onstep (Experimental): Participants in this group will have an inguinal hernia repair ad modum Onstep.
  Interventions: Procedure: Onstep
- Laparoscopic repair (Active Comparator): Participants in this group will receive an inguinal hernia repair by use of a laparoscopic approach.
  Interventions: Procedure: Laparoscopic repair

INTERVENTIONS:
Procedure: Onstep
  Arms: Onstep
Procedure: Laparoscopic repair
  Arms: Laparoscopic repair

SUMMARY:
The objective of this study is to evaluate chronic pain after inguinal hernia repair involving mesh placement with the Onstep-technique compared to mesh placement using a laparoscopic approach. The study hypothesis is that an even or smaller proportions of patients operated the Onstep technique will have chronic pain that impairs daily function.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnose of a primary groin hernia that requires surgical intervention.
* Eligible for procedure performed under general anesthesia.
* Eligible for both laparoscopic and Onstep procedure.

Exclusion Criteria:

* Not able to understand Danish/Swedish, written and spoken.
* Emergency procedures.
* Previous inguinal hernia on ipsilateral side.
* ASA score more than 3.
* Irreducible inguinoscrotal hernia.
* Local or systemic infection.
* Contralateral hernia being operated at the same time or planned operated during follow-up.
* Other abdominal hernias being operated at the same time or planned operated during follow-up.
* Previous surgery that has impaired the sensation in the groin area.
* BMI > 40 or < 20.
* Daily intake of alcohol >5 units, 1 unit = 12g pure alcohol.
* Known disease which impairs central or peripheral nerve function.
* Concurrent malignant disease.
* Impairment of cognitive function (e.g. dementia).
* Chronic pain that requires medication.
* Mental disorder that requires medication.

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2014-03; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with substantial pain related impairment of function | 6 month
  At the 6 month follow up, all participants will be asked to fill out questionnaires regarding pain. Questionnaire used will assess degree of pain and degree of impairment on daily function.
Early postoperative pain | 10 days
  Early postoperative pain, measured on postoperative day 1, 2, 3 and 10 on the VAS for pain and compared between groups.
Pain related impairment of function at 12 months | 12 months
  At the 12 months follow up, all participants will be asked to fill out questionnaires regarding pain. Questionnaire used will assess degree of pain and degree of impairment on daily function.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Rosenberg, Professor, Study Chair — University of Copenhagen, Herlev Hospital
Locations (1):
- Department of Surgery, Herlev Hospital, Herlev, Denmark

REFERENCES:
- [Derived] Andresen K, Burcharth J, Rosenberg J. ONSTEP versus laparoscopy for inguinal hernia repair: protocol for a randomised clinical trial. Dan Med J. 2015 Dec;62(12):A5169. PMID 26621399